CLINICAL TRIAL: NCT04847037
Title: Place of Connected Tools in the Follow-up of the Bariatric Patient: Can They Allow Rapid Management of Complications and Reduce Lost of Follow-up During Postoperative Period?
Brief Title: Place of Connected Tools in Bariatric Patients Follow-up.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Elsan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dr CARANDINA; 2019-A01371-56 (Other: ANSM)
Record Dates: First submitted 2021-04-14; First posted 2021-04-15 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Bariatric Surgery Candidate

STUDY DESIGN:
Intervention Model Description: This is a pilot, prospective, single-center, comparative, randomized, open-label study.
Masking Description: The experimental group which will use the connected tools will be compared with the control group according to the usual procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connected Tools (Experimental): For the experimental group, the postoperative procedure requires the use of personal connected tools: a smartphone, a digital tablet or a computer with internet connection. A scale and a connected watch will also be loaned to patients so that they can take the necessary measures. Before returning home, patients must be trained to take correct measures and inform them on the dedicated platform.
  Interventions: Procedure: Connected tools
- No Connected Tools (No Intervention): Patients randomized to the control group will be operated according to the same protocol as the experimental group. For them, there will be no home follow-up, so no special procedure to follow.

INTERVENTIONS:
Procedure: Connected tools — Use of connected tools in postoperative bariatric follow-up vs no use of connected tools.
  Arms: Connected Tools

SUMMARY:
The aim of this study is to assess the safety (in terms of post-operative complications) of the use of connected devices for the monitoring of patients operated on by longitudinal laparoscopic gastrectomy (LSG) and discharged 24 hours after surgery according to the protocol Enhanced Recovery After Surgery (ERAS).

DETAILED DESCRIPTION:
Connected devices, such as electronic scales and brachial cuffs used during the preoperative period, can help patients to self-control their weight and blood pressure and to better control certain risk factors for surgery. In addition, in order to reduce the number of deaths in the wards after surgery, connected devices have been designed to continuously monitor the vital parameters of patients. Subbe et al. recently showed that the use of wireless sensors to continuously monitor heart rate, respiratory rate, blood pressure and Oxygen Saturation by Pulse Oximetry (SpO2) reduced the number of cardiac arrests and mortality during hospitalization. Likewise, connected devices could potentially be used to monitor the patient directly at home and thus allow a faster discharge from the hospital without increasing the risks for the patient. At the current stage, there are no studies that have demonstrated the benefit of using the tools connected in postoperative follow-up in bariatric surgery.

Recently, thanks to the growth of experience and the application of the ERAS method, the postoperative stay at LSG has significantly decreased. Despite this, there are still very few centers that perform this operation in outpatient surgery or with a 24-hour hospital stay. This is probably due not only to a strict selection criteria, but also to the surgeon's concern to discharge the patient too early without medical supervision. In this context, the use of connected devices making it possible to monitor the patient directly at home and therefore theoretically continue a kind of medical surveillance could make it possible to increase the number of LSG performed in outpatient surgery. In addition, another advantage of this postoperative monitoring system is that it gives the patient a central role in the healing process after surgery. Thanks to devices and the Internet platform, the patient actively participates in his monitoring and remains in permanent contact with the surgical department. In this way, the feeling of fragility and loneliness that often feels the patient when he quickly returns home is reduced. Thus, compared to a small expense related to the purchase of devices, this would result in a significant reduction in hospital costs for the health system. The more important limitation of this procedure remains the degree of familiarity of the patient with the connected tools, and therefore will not necessarily be applicable to the entire population of obese patients without the risks of having a significant lack of follow-up during the first postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a BMI between 35 and 40 and comorbidity (type II diabetes, arterial hypertension, sleep apnea syndrome, dyslipidemia, fatty liver disease, arthropathy linked to overweight) related to obesity
* Patients with a BMI greater than 40 with or without comorbidity
* Patients affiliated to the social security scheme, with or without mutual health insurance
* Collection of signed informed consent
* Patients with one of the following sets of tools:

  * Computer tablet and computer with an internet connection
  * Computer tablet and smartphone with an internet connection
  * Smartphone and computer with an internet connection
* Patients without a history of bariatric surgery
* Patients with surgical indication for a sleeve gastrectomy

Exclusion Criteria:

* Patients who have had obesity surgery
* Patients who have the indication but want another surgery such as the sleeve
* Patients who do not have an internet connection and / or an email address
* Patients with a BMI less than 35
* Patients with a major contraindication to surgery and / or American Society of Anesthesiologists (ASA) 4
* Patients without social security
* Patients refusing to sign consent
* Patients living abroad and / or living more than two hours from the hospital
* Minors or patients over 70 years old

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2022-04-05 (Actual); Study Completion 2025-03-05 (Estimated)

PRIMARY OUTCOMES:
Complication Rate measured at 30 days. | 30 days after gastrectomy intervention.
  The complication rate will be compared in the both treatment groups.

SECONDARY OUTCOMES:
Rate of lost to follow-up at 3 years. | 3 years after gastrectomy intervention/
  The rate of lost to follow-up will be compared in the both treatment groups.
Change in the lost to follow-up rate at 1 year. | 1 year after gastrectomy intervention.
  In order to evaluate the evolution of the lost to follow-up, the change from baseline will be analyzed between the two treatment groups.
Change in the lost to follow-up rate at 2 years. | 2 years after gastrectomy intervention.
  In order to evaluate the evolution of the lost to follow-up, the change from baseline will be analyzed between the two treatment groups.
Change in the loss to follow-up rate at 3 years. | 3 years after gastrectomy intervention.
  In order to evaluate the evolution of the lost to follow-up, the change from baseline will be analyzed between the two treatment groups.
Patient satisfaction regarding the use of tools. | 15 days after gastrectomy intervention.
  A satisfaction questionnaire adapted to the study will be presented to patients in order to evaluate the satisfaction of tools' using, only for experimental group.
Quality of life assessment at 3 months. | 3 months after gastrectomy intervention.
  The BAROS quality of life questionnaire will be presented to patients in order to evaluate the quality of life.
Quality of life assessment at 6 months. | 6 months after gastrectomy intervention.
  The BAROS quality of life questionnaire will be presented to patients in order to evaluate the quality of life.
Quality of life assessment at 12 months. | 12 months after gastrectomy intervention.
  The BAROS quality of life questionnaire will be presented to patients in order to evaluate the quality of life.
Post-operative complications at 3 months | 3 months after gastrectomy intervention.
  The post-operative complications will be collected in both groups to evaluate the complication rate.
Post-operative complications at 6 months | 6 months after gastrectomy intervention.
  The post-operative complications will be collected in both groups to evaluate the complication rate.
Post-operative complications at 12 months | 12 months after gastrectomy intervention.
  The post-operative complications will be collected in both groups to evaluate the complication rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Chirurgical d'Obesité, Toulon, France

REFERENCES:
- [Background] Stevens GA, Singh GM, Lu Y, Danaei G, Lin JK, Finucane MM, Bahalim AN, McIntire RK, Gutierrez HR, Cowan M, Paciorek CJ, Farzadfar F, Riley L, Ezzati M; Global Burden of Metabolic Risk Factors of Chronic Diseases Collaborating Group (Body Mass Index). National, regional, and global trends in adult overweight and obesity prevalences. Popul Health Metr. 2012 Nov 20;10(1):22. doi: 10.1186/1478-7954-10-22. PMID 23167948
- [Background] Bult MJ, van Dalen T, Muller AF. Surgical treatment of obesity. Eur J Endocrinol. 2008 Feb;158(2):135-45. doi: 10.1530/EJE-07-0145. PMID 18230819
- [Background] Nguyen NT, Nguyen B, Gebhart A, Hohmann S. Changes in the makeup of bariatric surgery: a national increase in use of laparoscopic sleeve gastrectomy. J Am Coll Surg. 2013 Feb;216(2):252-7. doi: 10.1016/j.jamcollsurg.2012.10.003. Epub 2012 Nov 21. PMID 23177371
- [Background] Simonelli V, Goergen M, Orlando GG, Arru L, Zolotas CA, Geeroms M, Poulain V, Azagra JS. Fast-Track in Bariatric and Metabolic Surgery: Feasibility and Cost Analysis Through a Matched-Cohort Study in a Single Centre. Obes Surg. 2016 Aug;26(8):1970-7. doi: 10.1007/s11695-016-2255-4. PMID 27272321
- [Background] Malczak P, Pisarska M, Piotr M, Wysocki M, Budzynski A, Pedziwiatr M. Enhanced Recovery after Bariatric Surgery: Systematic Review and Meta-Analysis. Obes Surg. 2017 Jan;27(1):226-235. doi: 10.1007/s11695-016-2438-z. PMID 27817086
- [Background] Khorgami Z, Petrosky JA, Andalib A, Aminian A, Schauer PR, Brethauer SA. Fast track bariatric surgery: safety of discharge on the first postoperative day after bariatric surgery. Surg Obes Relat Dis. 2017 Feb;13(2):273-280. doi: 10.1016/j.soard.2016.01.034. Epub 2016 Feb 2. PMID 27986577
- [Background] Rebibo L, Dhahri A, Badaoui R, Dupont H, Regimbeau JM. Laparoscopic sleeve gastrectomy as day-case surgery (without overnight hospitalization). Surg Obes Relat Dis. 2015 Mar-Apr;11(2):335-42. doi: 10.1016/j.soard.2014.08.017. Epub 2014 Sep 16. PMID 25614354
- [Background] Varadhan KK, Neal KR, Dejong CH, Fearon KC, Ljungqvist O, Lobo DN. The enhanced recovery after surgery (ERAS) pathway for patients undergoing major elective open colorectal surgery: a meta-analysis of randomized controlled trials. Clin Nutr. 2010 Aug;29(4):434-40. doi: 10.1016/j.clnu.2010.01.004. Epub 2010 Jan 29. PMID 20116145
- [Background] Spanjersberg WR, Reurings J, Keus F, van Laarhoven CJ. Fast track surgery versus conventional recovery strategies for colorectal surgery. Cochrane Database Syst Rev. 2011 Feb 16;(2):CD007635. doi: 10.1002/14651858.CD007635.pub2. PMID 21328298
- [Background] Berg K, Arestedt K, Kjellgren K. Postoperative recovery from the perspective of day surgery patients: a phenomenographic study. Int J Nurs Stud. 2013 Dec;50(12):1630-8. doi: 10.1016/j.ijnurstu.2013.05.002. Epub 2013 May 30. PMID 23726224
- [Background] Svensson M, Nilsson U, Svantesson M. Patients' experience of mood while waiting for day surgery. J Clin Nurs. 2016 Sep;25(17-18):2600-8. doi: 10.1111/jocn.13304. Epub 2016 Jun 27. PMID 27349201
- [Background] Michard F. Smartphones and e-tablets in perioperative medicine. Korean J Anesthesiol. 2017 Oct;70(5):493-499. doi: 10.4097/kjae.2017.70.5.493. Epub 2017 Sep 28. PMID 29046768
- [Background] Jaensson M, Dahlberg K, Eriksson M, Nilsson U. Evaluation of postoperative recovery in day surgery patients using a mobile phone application: a multicentre randomized trial. Br J Anaesth. 2017 Nov 1;119(5):1030-1038. doi: 10.1093/bja/aex331. PMID 29077818
- [Background] Topol EJ. Transforming medicine via digital innovation. Sci Transl Med. 2010 Jan 27;2(16):16cm4. doi: 10.1126/scitranslmed.3000484. PMID 20371472
- [Background] Noar SM, Black HG, Pierce LB. Efficacy of computer technology-based HIV prevention interventions: a meta-analysis. AIDS. 2009 Jan 2;23(1):107-15. doi: 10.1097/QAD.0b013e32831c5500. PMID 19050392
- [Background] Whittaker R, McRobbie H, Bullen C, Rodgers A, Gu Y. Mobile phone-based interventions for smoking cessation. Cochrane Database Syst Rev. 2016 Apr 10;4(4):CD006611. doi: 10.1002/14651858.CD006611.pub4. PMID 27060875
- [Background] Oosterveen E, Tzelepis F, Ashton L, Hutchesson MJ. A systematic review of eHealth behavioral interventions targeting smoking, nutrition, alcohol, physical activity and/or obesity for young adults. Prev Med. 2017 Jun;99:197-206. doi: 10.1016/j.ypmed.2017.01.009. Epub 2017 Jan 25. PMID 28130046
- [Background] Broekhuizen K, Kroeze W, van Poppel MN, Oenema A, Brug J. A systematic review of randomized controlled trials on the effectiveness of computer-tailored physical activity and dietary behavior promotion programs: an update. Ann Behav Med. 2012 Oct;44(2):259-86. doi: 10.1007/s12160-012-9384-3. PMID 22767052
- [Background] Stephenson A, McDonough SM, Murphy MH, Nugent CD, Mair JL. Using computer, mobile and wearable technology enhanced interventions to reduce sedentary behaviour: a systematic review and meta-analysis. Int J Behav Nutr Phys Act. 2017 Aug 11;14(1):105. doi: 10.1186/s12966-017-0561-4. PMID 28800736
- [Background] Subbe CP, Duller B, Bellomo R. Effect of an automated notification system for deteriorating ward patients on clinical outcomes. Crit Care. 2017 Mar 14;21(1):52. doi: 10.1186/s13054-017-1635-z. PMID 28288655
- [Background] Angrisani L, Santonicola A, Iovino P, Vitiello A, Higa K, Himpens J, Buchwald H, Scopinaro N. IFSO Worldwide Survey 2016: Primary, Endoluminal, and Revisional Procedures. Obes Surg. 2018 Dec;28(12):3783-3794. doi: 10.1007/s11695-018-3450-2. PMID 30121858
- [Background] Akkary E, Duffy A, Bell R. Deciphering the sleeve: technique, indications, efficacy, and safety of sleeve gastrectomy. Obes Surg. 2008 Oct;18(10):1323-9. doi: 10.1007/s11695-008-9551-6. Epub 2008 Jun 6. PMID 18535867
- [Background] Nocca D, Krawczykowsky D, Bomans B, Noel P, Picot MC, Blanc PM, de Seguin de Hons C, Millat B, Gagner M, Monnier L, Fabre JM. A prospective multicenter study of 163 sleeve gastrectomies: results at 1 and 2 years. Obes Surg. 2008 May;18(5):560-5. doi: 10.1007/s11695-007-9288-7. PMID 18317859
- [Background] Lalor PF, Tucker ON, Szomstein S, Rosenthal RJ. Complications after laparoscopic sleeve gastrectomy. Surg Obes Relat Dis. 2008 Jan-Feb;4(1):33-8. doi: 10.1016/j.soard.2007.08.015. Epub 2007 Nov 5. PMID 17981515
- [Background] Sethi M, Patel K, Zagzag J, Parikh M, Saunders J, Ude-Welcome A, Somoza E, Schwack B, Kurian M, Fielding G, Ren-Fielding C. Thirty-Day Readmission After Laparoscopic Sleeve Gastrectomy-a Predictable Event? J Gastrointest Surg. 2016 Feb;20(2):244-52. doi: 10.1007/s11605-015-2978-x. PMID 26487330
- [Background] Jonsson A, Lin E, Patel L, Patel AD, Stetler JL, Prayor-Patterson H, Singh A, Srinivasan JK, Sweeney JF, Davis SS Jr. Barriers to Enhanced Recovery after Surgery after Laparoscopic Sleeve Gastrectomy. J Am Coll Surg. 2018 Apr;226(4):605-613. doi: 10.1016/j.jamcollsurg.2017.12.028. Epub 2018 Jan 5. PMID 29309941
- [Background] Lalezari S, Musielak MC, Broun LA, Curry TW. Laparoscopic sleeve gastrectomy as a viable option for an ambulatory surgical procedure: our 52-month experience. Surg Obes Relat Dis. 2018 Jun;14(6):748-750. doi: 10.1016/j.soard.2018.02.015. Epub 2018 Feb 17. PMID 29567060
- [Background] te Riele WW, Boerma D, Wiezer MJ, Borel Rinkes IH, van Ramshorst B. Long-term results of laparoscopic adjustable gastric banding in patients lost to follow-up. Br J Surg. 2010 Oct;97(10):1535-40. doi: 10.1002/bjs.7130. PMID 20564686
- [Background] Althoff T, White RW, Horvitz E. Influence of Pokemon Go on Physical Activity: Study and Implications. J Med Internet Res. 2016 Dec 6;18(12):e315. doi: 10.2196/jmir.6759. PMID 27923778
- [Background] Thorell A, MacCormick AD, Awad S, Reynolds N, Roulin D, Demartines N, Vignaud M, Alvarez A, Singh PM, Lobo DN. Guidelines for Perioperative Care in Bariatric Surgery: Enhanced Recovery After Surgery (ERAS) Society Recommendations. World J Surg. 2016 Sep;40(9):2065-83. doi: 10.1007/s00268-016-3492-3. PMID 26943657
- [Background] Moorehead MK, Ardelt-Gattinger E, Lechner H, Oria HE. The validation of the Moorehead-Ardelt Quality of Life Questionnaire II. Obes Surg. 2003 Oct;13(5):684-92. doi: 10.1381/096089203322509237. PMID 14627461
- [Background] Nini E, Slim K, Scesa JL, Chipponi J. [Evaluation of laparoscopic bariatric surgery using the BAROS score]. Ann Chir. 2002 Feb;127(2):107-14. doi: 10.1016/s0003-3944(01)00688-5. French. PMID 11885369